CLINICAL TRIAL: NCT00813787
Title: Investigation Into the Differentiation of Tumour and Healthy Brain Tissue Using a Specialized MRI Technique Called Multiexponential T2 Component Analysis
Brief Title: Investigation Into the Differentiation of Tumour and Healthy Brain Tissue Using Multi-exponential T2 Components
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: CNS-24534
Record Dates: First submitted 2008-12-19; First posted 2008-12-23 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-10

CONDITIONS: Glioma
Keywords: Magnetic Resonance Imaging; Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- A. glioma: A. glioma population
- B. Normal brain: B. Normal brain

SUMMARY:
The purpose of this study is to see if a specialized imaging technique using MRI called multi-exponential T2 component analysis can reliably differentiate between normal brain and brain tumour.

DETAILED DESCRIPTION:
Existing methods of contouring tumours for radiation therapy involve manual interpretations of qualitative diagnostic images. These methods, being qualitative, do not offer a consistent and reproducible platform for contouring, making it difficult to evaluate the effects of contouring choices on treatment outcome. T2 component analysis in MRI has the potential to offer a quantitive basis for identifying tumor tissue- this potential is investigated in this pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Eighteen years of age or older
* Clinical subjects must have not yet begun radiation therapy
* Must have signed our study-specific consent form

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A. Any glioma patient who recieves treatment at our clinic (Cross Cancer Institute) who agrees to take part in the study.
  B. Any normal volunteer who agrees to take part in the study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2009-02; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
T2 characteristics of glioma tissue versus normal | Before radiotherapy treatment begins

CONTACTS AND LOCATIONS:
Overall Officials: Keith Wachowicz, PhD, Study Chair — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada